CLINICAL TRIAL: NCT02227875
Title: An Open-label, Randomized, Multi-center, Parallel Group Clinical Trial Comparing the Efficacy and Safety of Mylan's Insulin Glargine With Lantus® in Type 2 Diabetes Mellitus Patients
Brief Title: Non-inferiority Study to Compare the Efficacy and Safety of Mylan's Insulin Glargine With Lantus® in Type 2 Diabetes Mellitus Patients (INSTRIDE 2)
Acronym: INSTRIDE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYL-GAI-3002
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mylan's insulin Glargine (Experimental): receive Mylan's insulin Glargine
  Interventions: Drug: Mylan's insulin glargine
- Lantus® (Active Comparator): receive Lantus®
  Interventions: Drug: Lantus®

INTERVENTIONS:
Drug: Mylan's insulin glargine — Patients who are randomized to receive Mylan's insulin glargine during the comparative phase will receive the same dose as the dose of Lantus® received during the screening period. The recommended starting dose of Mylan's insulin glargine or Lantus®, in patients with T2DM who are not currently treated with insulin is 10 units (or 0.2 Units/kg) once daily, which should subsequently be adjusted every week if essential.
  Arms: Mylan's insulin Glargine
Drug: Lantus® — For patients who are randomized to receive Lantus® during the comparative phase the dose of Lantus® will be equal to the dose received during the screening period.
  Arms: Lantus®

SUMMARY:
To test whether Mylan's insulin glargine once daily is non-inferior to Lantus® once daily (both administered in combination with other anti-diabetic drugs) based on the change in HbA1c from baseline to 24 weeks

DETAILED DESCRIPTION:
This trial is a multi-center, open-label, randomized, parallel group trial in patients with T2DM comparing the efficacy and safety of Mylan's insulin glargine with that of Lantus®. Patients with an established diagnosis of T2DM per ADA 2014 criteria and who satisfy the selection criteria will be included in the trial. This will be followed by a 24-week randomized, comparative, parallel-assignment treatment period with Mylan's insulin glargine or Lantus® (in addition to other anti-diabetic drugs). After the treatment period, there will be a follow-up visit; 4 weeks after the patient has been put back on approved medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of T2DM per ADA 2014 criteria who also fulfill the following:

  * Diagnosis established 1 year prior to screening
  * Insulin-naïve OR
  * On Lantus® once daily at stable dose (±15% variation in dose) for at least 3 months prior to screening
* Body mass index (BMI) of 18.50 to 40.00 kg/m2 at screening (both values inclusive).
* Stable weight, with no more than 5 kg gain or loss, in the 3 months prior to screening; this information will be collected by patient interview during medical history.
* Hemoglobin ≥9.0 g/dL at screening
* Glycosylated hemoglobin (HbA1c) of <10.5% or between 7.5 to 10.5% for insulin naïve patients at screening.

Exclusion Criteria:

* History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analog preparations used in the trial, OR history of significant allergic drug reactions.
* History of use of animal insulin within the last 3 years, any insulin other than Lantus® within the last 3 months prior to screening, or use of biosimilar insulin glargine at any time prior to screening.
* Patients requiring basal-bolus insulin therapy or who in the opinion of the investigator require mealtime insulin in order to achieve glycemic control.
* Regular use of immune-modulator therapy in the 1 year prior to screening.
* History of ≥2 episodes of severe hypoglycemia within the 6 months before screening or history of hypoglycemia unawareness (a sample questionnaire is provided in Appendix I) as judged by the investigator.
* History of ≥1 episode of hyperglycemic hyperosmolar coma or emergency room visits for uncontrolled diabetes leading to hospitalization within the 6 months prior to screening.
* Serological evidence of human immunodeficiency virus (HIV), hepatitis B (HbSAg) or hepatitis C (HCVAb) antibodies at screening.
* History of drug or alcohol dependence or abuse during the 1 year prior to screening.
* Receipt of another investigational drug in the 3 months prior to screening (or as per local regulations), or if the screening visit is within 5 half-lives of another investigational drug (whichever is longer), or scheduled to receive another investigational drug during the current trial period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blevins, MD, Principal Investigator — Texas Diabetes & Endocrinology
Locations (112):
- United States (87):
  - Mylan Investigational Site, Chandler, Arizona
  - Mylan Investigational Site, Bell Gardens, California
  - Mylan Investigational Site, Fresno, California
  - Mylan Investigational Site, Greenbrae, California
  - Mylan Investigational Site, Long Beach, California
  - Mylan Investigational Site, Los Angeles, California
  - Mylan Investigational Site, Los Gatos, California
  - Mylan Investigational Site, Mission Hills, California
  - Mylan Investigational Site, National City, California
  - Mylan Investigational Site, Northridge, California
  - Mylan Investigational Site, Orange, California
  - Mylan Investigational Site, Palm Springs, California
  - Mylan Investigational Site, Spring Valley, California
  - Mylan Investigational Site, Tustin, California
  - Mylan Investigational Site, Walnut Creek, California
  - Mylan Investigational Site, West Hills, California
  - Mylan Investigational Site, Bradenton, Florida
  - Mylan Investigational Site, Cooper City, Florida
  - Mylan Investigational Site, Hialeah, Florida
  - Mylan Investigational Site, Miami, Florida
  - Mylan Investigational Site, New Port Richey, Florida
  - Mylan Investigational Site, Palm Harbor, Florida
  - Mylan Investigational Site, Pembroke Pines, Florida
  - Mylan Investigational Site, Port Charlotte, Florida
  - Mylan Investigational Site, West Palm Beach, Florida
  - Mylan Investigational Site, Winter Haven, Florida
  - Mylan Investigational Site, Columbus, Georgia
  - Mylan Investigational Site, Gainesville, Georgia
  - Mylan Investigational Site, Honolulu, Hawaii
  - Mylan Investigational Site, Idaho Falls, Idaho
  - Mylan Investigational Site, Chicago, Illinois
  - Mylan Investigational Site, Crystal Lake, Illinois
  - Mylan Investigational Site, Springfield, Illinois
  - Mylan Investigational Site, Anderson, Indiana
  - Mylan Investigational Site, Council Bluffs, Iowa
  - Mylan Investigational Site, Des Moines, Iowa
  - Mylan Investigational Site, Augusta, Kansas
  - Mylan Investigational Site, Topeka, Kansas
  - Mylan Investigational Site, Wichita, Kansas
  - Mylan Investigational Site, Crestview Hills, Kentucky
  - Mylan Investigational Site, Lexington, Kentucky
  - Mylan Investigational Site, Waltham, Massachusetts
  - Mylan Investigational Site, Kansas City, Missouri
  - Mylan Investigational Site, St Louis, Missouri
  - Mylan Investigational Site, Billings, Montana
  - Mylan Investigational Site, Lincoln, Nebraska
  - Mylan Investigational Site, Omaha, Nebraska
  - Mylan Investigational Site, Las Vegas, Nevada
  - Mylan Investigational Site, Nashua, New Hampshire
  - Mylan Investigational Site, Albany, New York
  - Mylan Investigational Site, Hartsdale, New York
  - Mylan Investigational Site, Smithtown, New York
  - Mylan Investigational Site, Staten Island, New York
  - Mylan Investigational Site, Asheville, North Carolina
  - Mylan Investigational Site, Burlington, North Carolina
  - Mylan Investigational Site, Cary, North Carolina
  - Mylan Investigational Site, Greensboro, North Carolina
  - Mylan Investigational Site, Greenville, North Carolina
  - Mylan Investigational Site, Hickory, North Carolina
  - Mylan Investigational Site, Morehead City, North Carolina
  - Mylan Investigational Site, Wilmington, North Carolina
  - Mylan Investigational Site, Cincinnati, Ohio
  - Mylan Investigational Site, Cleveland, Ohio
  - Mylan Investigational Site, Columbus, Ohio
  - Mylan Investigational Site, Bend, Oregon
  - Mylan Investigational Site, Charleston, South Carolina
  - Mylan Investigational Site, Greer, South Carolina
  - Mylan Investigational Site, Bristol, Tennessee
  - Mylan Investigational Site, Kingsport, Tennessee
  - Mylan Investigational Site, Memphis, Tennessee
  - Mylan Investigational Site, Austin, Texas
  - Mylan Investigational Site, Corpus Christi, Texas
  - Mylan Investigational Site, Dallas, Texas
  - Mylan Investigational Site, El Paso, Texas
  - Mylan Investigational Site, Houston, Texas
  - Mylan Investigational Site, McKinney, Texas
  - Mylan Investigational Site, Round Rock, Texas
  - Mylan Investigational Site, San Antonio, Texas
  - Mylan Investigational Site, Spring, Texas
  - Mylan Investigational Site, Victoria, Texas
  - Mylan Investigational Site, Ogden, Utah
  - Mylan Investigational Site, Salt Lake City, Utah
  - Mylan Investigational Site, South Jordan, Utah
  - Mylan Investigational Site, Chesapeake, Virginia
  - Mylan Investigational Site, Manassas, Virginia
  - Mylan Investigational Site, Tacoma, Washington
  - Mylan Investigational Site, Vancouver, Washington
- Jordan (2):
  - Mylan Investigational Site, Amman
  - Mylan Investigational Site, Irbid
- Slovakia (13):
  - Mylan Investigational Site, Banská Bystrica
  - Mylan Investigational Site, Bardejov
  - Mylan Investigational Site, Bratislava
  - Mylan Investigational Site, Dolný Kubín
  - Mylan Investigational Site, Košice
  - Mylan Investigational Site, Levice
  - Mylan Investigational Site, Sabinov
  - Mylan Investigational Site, Stropkov
  - Mylan Investigational Site, Šahy
  - Mylan Investigational Site, Štúrovo
  - Mylan Investigational Site, Trebišov
  - Mylan Investigational Site, Trenčín
  - Mylan Investigational Site, Žilina
- South Africa (5):
  - Mylan Investigational Site, Johannesburg, Gauteng
  - Mylan Investigational Site, Durban, KwaZulu-Natal
  - Mylan Investigational Site, Cape Town, Western Cape
  - Mylan Investigational Site, Worcester, Western Cape
  - Mylan Investigational Site, Bloemfontein
- South Korea (3):
  - Mylan Investigational Site, Seoul, Gyeonggi-do
  - Mylan Investigational Site, Suwon, Gyeonggi-do
  - Mylan Investigational Site, Seoul
- Taiwan (2):
  - Mylan Investigational Site, Kaohsiung City
  - Mylan Investigational Site, Taipei

REFERENCES:
- [Derived] Sun B, Sengupta N, Rao A, Donnelly C, Waichale V, Roy AS, Ramaswamy S, Pathak D, Bowsher RR, Raiter Y, Aubonnet P, Barve A. Similar immunogenicity profiles between the proposed biosimilar MYL-1501D and reference insulin glargine in patients with diabetes mellitus: the phase 3 INSTRIDE 1 and INSTRIDE 2 studies. BMC Endocr Disord. 2021 Jun 26;21(1):129. doi: 10.1186/s12902-021-00797-4. PMID 34174848

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mylan's Insulin Glargine | Lantus®
Started | 277 | 283
Completed | 240 | 250
Not Completed | 37 | 33
Not completed — Protocol Violation | 10 | 7
Not completed — Other | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 12 | 13
Not completed — Lost to Follow-up | 10 | 10

BASELINE CHARACTERISTICS:
Population: Recruitment details:
  * Gender: male or female;
  * Age: 18-65 years, inclusive;
  * Body mass index (BMI): 18.5-40.0 kg/m2, inclusive
Groups:
- Total: Total of all reporting groups
Arm/Group | Mylan's Insulin Glargine | Lantus® | Total
Number analyzed (Participants) | 277 | 283 | 560
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 267 | 267 | 534
  >=65 years | 10 | 16 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7.91) | 55.1 (7.5) | 55.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 118 | 248
  Male | 147 | 165 | 312
Region of Enrollment [Number; unit: participants]
  South Korea | 3 | 4 | 7
  United States | 225 | 228 | 453
  Taiwan | 1 | 0 | 1
  South Africa | 12 | 15 | 27
  Slovakia | 34 | 33 | 67
  Jordan | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to 24 Weeks
Time Frame: 24 weeks
Population: Intent-to-Treat Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 274 | 278
percent | -0.6 [-0.779 to -0.414] | -0.66 [-0.837 to -0.475]
Statistical Analysis 1: Comparison: Mylan's Insulin Glargine vs Lantus®; Test type: Non-Inferiority — Mixed-Effect Model for Repeated Measures; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.098 to 0.218], Standard Error of Mean 0.08

2. Secondary Outcome: Rate of Hypoglycemic Events Per 30 Days
Description: The change from baseline at 12 and 24 weeks is reported
Time Frame: Baseline and up to 24 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Episodes/30 Days
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 276 | 282
Episodes/30 Days
  week 12 | 0.341 (1.8963) | 0.24 (2.0551)
  week 24 | -0.057 (0.919) | -0.102 (1.6791)

3. Secondary Outcome: Hypoglycemia Occurrence
Description: Overall hypoglycemic incidence during treatment period
Time Frame: 24 weeks
Population: Safety Population
Measure: Number; unit: number of events
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 276 | 282
number of events
  Any hypoglycemic event | 130 | 136
  Severe Hypoglycemia | 0 | 1
  Documented Symptomatic Hypoglycemia | 75 | 76
  Asymptomatic Hypoglycemia | 85 | 92
  Probable Symptomatic Hypoglycemia | 7 | 4
  Relative Hypoglycemia | 20 | 11
  Unknown | 29 | 25

4. Secondary Outcome: Change in Total Insulin Antibody Percent Binding for Mylan's Insulin Glargine Assay Over Time
Description: Comparison of change from Baseline in Immunogenicity
Time Frame: Week 12 and week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of specific binding (SB)
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 276 | 282
percentage of specific binding (SB)
  week 12 | 1.9238 (12.54369) | 0.6585 (8.05473)
  week 24 | 1.7802 (9.64745) | 0.7838 (8.15086)

5. Secondary Outcome: Change in Total Insulin Antibody Percent Binding for Lantus Assay Over Time
Description: Comparison of change from Baseline in Immunogenicity
Time Frame: week 12 and week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of SB
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 276 | 282
percentage of SB
  week 12 | 1.787 (11.67578) | 0.6462 (7.56375)
  week 24 | 1.6866 (9.57132) | 0.8212 (8.1084)

6. Secondary Outcome: Change in Cross-Reactive Insulin Antibody Percent Binding for Mylan's Insulin Glargine Assay Over Time
Description: Comparison of change from Baseline in Immunogenicity
Time Frame: week 12 and week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of SB
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 276 | 282
percentage of SB
  week 12 | 1.7488 (11.68129) | 0.5116 (7.25175)
  week 24 | 1.6301 (9.11098) | 0.7524 (7.93317)

7. Secondary Outcome: Change in Cross-Reactive Insulin Antibody Percent Binding for Lantus Assay Over Time
Description: Comparison of change from Baseline in Immunogenicity
Time Frame: Week 12 and week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of SB
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 276 | 282
percentage of SB
  week 12 | 1.5994 (10.64782) | 0.5014 (6.72058)
  week 24 | 1.5648 (9.04243) | 0.8361 (7.96308)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Mylan's Insulin Glargine | Lantus®
All-Cause Mortality (participants affected / at risk) | 0/276 | 0/282
Serious Adverse Events (participants affected / at risk) | 8/276 | 9/282
Other Adverse Events (participants affected / at risk) | 177/276 | 164/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mylan's Insulin Glargine (N=276) | Lantus® (N=282)
Helicobacter test positive (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mylan's Insulin Glargine (N=276) | Lantus® (N=282)
Hypertension (Vascular disorders) | 6 (6) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 4 (4) | 2 (2)
Injection site pain (General disorders) | 3 (4) | 2 (3)
Oedema peripheral (General disorders) | 2 (2) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Lipase increased (Investigations) | 4 (4) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (10)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 10 (11)
Tremor (Nervous system disorders) | 6 (9) | 1 (3)
Dizziness (Nervous system disorders) | 4 (4) | 7 (8)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (10)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 75 (330) | 66 (282)
Upper respiratory tract infection (Infections and infestations) | 17 (19) | 15 (15)
Urinary tract infection (Infections and infestations) | 12 (13) | 8 (8)
Nasopharyngitis (Infections and infestations) | 10 (11) | 13 (14)
Sinusitis (Infections and infestations) | 8 (9) | 4 (5)
Influenza (Infections and infestations) | 6 (7) | 3 (3)
Bronchitis (Infections and infestations) | 5 (5) | 7 (7)
Gastroenteritis (Infections and infestations) | 5 (5) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days